CLINICAL TRIAL: NCT03179566
Title: Safe Opioid Disposal After Surgery Trial
Brief Title: Pain and Medication Use Following Surgery
Acronym: SODAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other)
Responsible Party: Principal Investigator, Chad Brummett, Associate Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00129418; MA-2017 (Other Grant/Funding Number: Michigan Department of Health and Human Services)
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Opioid Use
Keywords: drug disposal

STUDY DESIGN:
Intervention Model Description: A run-in period will precede the randomization sequence. Individuals will be randomized to one of two groups based on the day of their surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): For the first two weeks, there will be no intervention or changes to the usual discharge instructions
- Information Sheet (Active Comparator): At discharge, patients will receive an informational sheet detailing options for safe drug disposal
  Interventions: Behavioral: Information Sheet
- Deterra Drug Deactivation System (Active Comparator): At discharge, patients will receive a Deterra Drug Deactivation System.
  Interventions: Behavioral: Information Sheet; Behavioral: Deterra Drug Deactivation System

INTERVENTIONS:
Behavioral: Information Sheet — Patients will receive an informational sheet about how to dispose of leftover opioid medication during discharge. Nurses will provide this information sheet and a brief, scripted description of its use and importance of safe disposal at the time of discharge following surgery.
  Arms: Deterra Drug Deactivation System; Information Sheet
Behavioral: Deterra Drug Deactivation System — This system is a pouch that deactivates prescription drugs, rendering them ineffective for misuse and safe for regular garbage disposal. It uses a patented activated carbon technology to deactivate drugs, including pills, liquids, and patches, and has been found to be 99% percent effective in studies funded by the National Institute of Drug Abuse (NIDA). Additionally, the pouches are made from environmentally friendly materials and contain active ingredients that are considered non-toxic and pose minimal risk, according to their MSDS. Nurses will provide the Deterra bag and a brief, scripted description of its use and importance of safe disposal at the time of discharge following surgery.
  Arms: Deterra Drug Deactivation System

SUMMARY:
Patients will be randomized to one of two interventions intended to facilitate safe disposal of opioids after cessation following surgery. For pragmatic reasons, participants will be randomized by day to either the information sheet or the disposal bag using a block randomization schedule. To ensuring adequate sample size, patients will be enrolled for a ~4-week period following the 2-week usual care run in period. In the event that the sample size estimate has not been reached after the 4-week intervention period, additional patients will be enrolled accordingly.

DETAILED DESCRIPTION:
The lack of evidence-based guidelines for postoperative opioid prescribing has contributed to a surplus of opioid pills within our patients' homes and communities, increasing the potential for diversion and nonmedical use. A recent study suggests that for outpatient general surgery procedures, roughly 72% of prescribed opioids go unused. Current opioid disposal options are limited to DEA-authorized opioid collectors, including select law enforcement agencies, pharmacies, or organized pill drop events, and many patients remain unaware of these avenues. Several studies have found that few patients have knowledge about opioid disposal options and even fewer dispose of their unconsumed opioids.

Unconsumed opioids pose a diversion risk. In the 2011 National Survey on Drug Use and Health, 70.8% of those who used a prescription medication non-medically obtained the medication from a friend or relative, with or without their knowledge. Additionally, nonmedical prescription opioid use is a common pathway to heroin use. Importantly, over 80% of young intravenous drug users report initiation of prescription opioid misuse prior to heroin.

Considering that 40% of the prescriptions written by surgeons are for opioids and patients frequently have excess opioids and limited options for and/or knowledge of opioid disposal, the present study will provide patients with information and novel options for opioid disposal as part of the surgical care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgery at Michigan Medicine's East Ann Arbor Ambulatory Surgery & Medical Procedures Center

Exclusion Criteria:

* Unable to speak English
* Inability to understand or complete the surveys
* Other conditions that preclude meaningful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Drug disposal | 4 weeks post-surgery
  Patient-reported disposal of left-over opioid medications in any manner

SECONDARY OUTCOMES:
Opioid disposal technique | 4 weeks post-surgery
  Patient-reported technique for disposal of left-over opioid medications specifically assessing for safe disposal using recommended disposal methods

CONTACTS AND LOCATIONS:
Overall Officials: Chad Brummett, MD, Principal Investigator — Michigan Medicine, Department of Anesthesiology
Locations (1):
- East Ann Arbor Ambulatory Surgery & Medical Procedures Center - Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudd RA, Aleshire N, Zibbell JE, Gladden RM. Increases in Drug and Opioid Overdose Deaths--United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2016 Jan 1;64(50-51):1378-82. doi: 10.15585/mmwr.mm6450a3. PMID 26720857
- [Background] Levy B, Paulozzi L, Mack KA, Jones CM. Trends in Opioid Analgesic-Prescribing Rates by Specialty, U.S., 2007-2012. Am J Prev Med. 2015 Sep;49(3):409-13. doi: 10.1016/j.amepre.2015.02.020. Epub 2015 Apr 18. PMID 25896191
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Background] Reddy A, de la Cruz M, Rodriguez EM, Thames J, Wu J, Chisholm G, Liu D, Frisbee-Hume S, Yennurajalingam S, Hui D, Cantu H, Marin A, Gayle V, Shinn N, Xu A, Williams J, Bruera E. Patterns of storage, use, and disposal of opioids among cancer outpatients. Oncologist. 2014 Jul;19(7):780-5. doi: 10.1634/theoncologist.2014-0071. Epub 2014 May 27. PMID 24868100
- [Background] Egan KL, Gregory E, Sparks M, Wolfson M. From dispensed to disposed: evaluating the effectiveness of disposal programs through a comparison with prescription drug monitoring program data. Am J Drug Alcohol Abuse. 2017 Jan;43(1):69-77. doi: 10.1080/00952990.2016.1240801. Epub 2016 Oct 31. PMID 27797283
- [Background] Tanabe P, Paice JA, Stancati J, Fleming M. How do emergency department patients store and dispose of opioids after discharge? A pilot study. J Emerg Nurs. 2012 May;38(3):273-9. doi: 10.1016/j.jen.2011.09.023. Epub 2011 Dec 26. PMID 22204885
- [Background] Lewis ET, Cucciare MA, Trafton JA. What do patients do with unused opioid medications? Clin J Pain. 2014 Aug;30(8):654-62. doi: 10.1097/01.ajp.0000435447.96642.f4. PMID 24281287
- [Background] McCabe SE, West BT, Boyd CJ. Leftover prescription opioids and nonmedical use among high school seniors: a multi-cohort national study. J Adolesc Health. 2013 Apr;52(4):480-5. doi: 10.1016/j.jadohealth.2012.08.007. Epub 2012 Nov 22. PMID 23298996
- [Background] Voepel-Lewis T, Wagner D, Tait AR. Leftover prescription opioids after minor procedures: an unwitting source for accidental overdose in children. JAMA Pediatr. 2015 May;169(5):497-8. doi: 10.1001/jamapediatrics.2014.3583. No abstract available. PMID 25798880
- [Background] Vaughn MG, Nelson EJ, Salas-Wright CP, Qian Z, Schootman M. Racial and ethnic trends and correlates of non-medical use of prescription opioids among adolescents in the United States 2004-2013. J Psychiatr Res. 2016 Feb;73:17-24. doi: 10.1016/j.jpsychires.2015.11.003. Epub 2015 Nov 11. PMID 26679761
- [Background] Boyd CJ, Esteban McCabe S, Teter CJ. Medical and nonmedical use of prescription pain medication by youth in a Detroit-area public school district. Drug Alcohol Depend. 2006 Jan 4;81(1):37-45. doi: 10.1016/j.drugalcdep.2005.05.017. Epub 2005 Jul 22. PMID 16040201
- [Background] Fortuna RJ, Robbins BW, Caiola E, Joynt M, Halterman JS. Prescribing of controlled medications to adolescents and young adults in the United States. Pediatrics. 2010 Dec;126(6):1108-16. doi: 10.1542/peds.2010-0791. Epub 2010 Nov 29. PMID 21115581
- [Background] Lankenau SE, Teti M, Silva K, Jackson Bloom J, Harocopos A, Treese M. Initiation into prescription opioid misuse amongst young injection drug users. Int J Drug Policy. 2012 Jan;23(1):37-44. doi: 10.1016/j.drugpo.2011.05.014. Epub 2011 Jun 20. PMID 21689917